CLINICAL TRIAL: NCT03266783
Title: Comparison of Bleeding Risk Between Rivaroxaban and Apixaban for the Treatment of Acute Venous Thromboembolism
Acronym: COBRRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COBRRA
Record Dates: First submitted 2017-08-10; First posted 2017-08-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban group (Active Comparator): 10 mg orally (PO), twice a day (BID) for 1 week, then 5 mg PO BID for 3 months of treatment
  Interventions: Drug: Apixaban
- Rivaroxaban group (Active Comparator): 15 mg orally (PO), twice a day (BID) for 3 weeks, then 20 mg PO once a day (OD) for 3 months of treatment
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Apixaban — Refer to Apixaban group
  Other Names: Eliquis
  Arms: Apixaban group
Drug: Rivaroxaban — Refer to Rivaroxaban group
  Other Names: Xarelto
  Arms: Rivaroxaban group

SUMMARY:
Apixaban and rivaroxaban have been compared to standard therapy for treatment of acute symptomatic venous thromboembolism (VTE) in randomized controlled trials (RCTs), and are both approved by Health Canada. No safety or efficacy data is available from direct head-to-head comparison of these two anticoagulants. Lawsuits in the United States over bleeding events, patient perceptions, and concerns with medication adherence are additional factors highlighting the importance of a comparison trial. This multi-center, pragmatic, prospective, randomized, open-label, blinded end-point (PROBE) trial aims to compare the safety of apixaban and rivaroxaban for the treatment of VTE.

DETAILED DESCRIPTION:
VTE is the third leading cause of mortality by cardiovascular disease. Standard treatment for acute VTE uses a combination of parenteral Low-Molecular-Weight Heparin (LMWH) and oral vitamin K antagonists (VKA) for 3 months, and carries significant bleeding risk. The major and/or clinically-relevant non-major bleeding (CRNMB) event rate is reported between 8.1-9.7% during initial treatment. This treatment is burdensome owing to subcutaneous injections, drug interactions, and laboratory monitoring. Direct oral anticoagulants (DOACs) are simpler to use and do not require laboratory monitoring.

Rivaroxaban and apixaban are two DOACs targeting Factor Xa. Each DOAC was separately proven effective and safe when compared to standard treatment. Comparison of the bleeding rates between studies would favour use of apixaban over rivaroxaban; however, trial limitations and lack of direct comparison between these two agents makes it impossible to draw firm conclusions. This represents a dilemma in clinical practice because the absence of convincing differences in safety has led to genuine uncertainty about which DOAC has the best risk-to-benefit ratio.

To address these limitations, a head-to-head randomized controlled trial (RCT) is needed to determine the safety (i.e. bleeding risk) of twice daily apixaban over once daily rivaroxaban during the first 3 months of acute VTE treatment. Eligibility criteria will be less stringent than the COBRRA pilot study and reflect real-world patients. Cost-effective analysis of apixaban twice daily compared to rivaroxaban once daily will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed newly diagnosed symptomatic acute venous thromboembolism (VTE) [proximal lower extremity deep vein thrombosis (DVT) or segmental or greater pulmonary embolism (PE)]
* Age ≥ 18 years old
* Informed consent obtained

Exclusion Criteria:

* Have received > 72 hours of therapeutic anticoagulation
* Creatinine clearance < 30 ml/min calculated with the Cockcroft-Gault formula
* Any contraindication for anticoagulation with apixaban or rivaroxaban as determined by the treating physician such as, but not limited to:

  * active bleeding,
  * active malignancy, defined as a) diagnosed with cancer within the past 6 months; or b) recurrent, regionally advanced or metastatic disease; or c) currently receiving treatment or have received any treatment for cancer during the 6 months prior to randomization; or d) a hematologic malignancy not in complete remission,
  * weight > 120 kg,
  * liver disease (Child-Pugh Class B or C),
  * use of contraindicated medications
  * another indication for long-term anticoagulation (e.g. atrial fibrillation)
  * pregnant (note below) or breastfeeding (Note: as reported by the patient or a pregnancy test will be ordered at the discretion of the treating physician for women of childbearing potential as per standard of care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2760 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
The rate of adjudicated clinically relevant bleeding (CRB) events | For the duration of the study: 3 months
  CRB events are defined as the composite of major bleeding (MB) events and clinically relevant non-major bleeding (CRNMB) events.

SECONDARY OUTCOMES:
Adjudicated Major Bleeding events | For the duration of the study: 3 months
  Major bleeding will be defined as fatal bleeding, and/or, Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in hemoglobin of ≥20 g/L, or leading to transfusion of ≥2 units of whole blood or red cells.
Adjudicated Clinically Relevant Non-Major Bleeding events | For the duration of the study: 3 months
  Clinically relevant non-major bleeding will be defined as any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:
  * Requiring medical intervention by a healthcare professional
  * Leading to hospitalization or increased level of care
  * Prompting a face to face (i.e., not just a telephone or electronic communication) evaluation
Adjudicated recurrent VTE events | For the duration of the study: 3 months
  Recurrent VTE will be confirmed with investigational reports including clinic notes, D-dimer results and imaging as per standard of care. Recurrent DVT will be confirmed by compression ultrasound revealing a new (compared to baseline/index ultrasound) area of non-compressibility in the popliteal vein or more proximal vein, or venography demonstrating a constant intraluminal filling defect in the popliteal vein or more proximal veins. Recurrent PE will be diagnosed if the V/Q scan is non-normal and a new unmatched segmental or greater perfusion defect is documented, or an intraluminal filling defect is seen on CTPA in a segmental or greater vessel that was previously free of thrombus, or pulmonary angiography demonstrating a constant intraluminal filling defect or a cutoff of a vessel >2.5 mm in diameter will be considered diagnostic for PE.
Adjudicated VTE-related deaths | For the duration of the study: 3 months
  VTE-related death (fatal PE or unexplained deaths) will be confirmed using death certificates and/or autopsy findings.
All-cause mortality | For the duration of the study: 3 months
  Using a binary outcome of an event or no event (Individual rates of death related to VTE, bleeding or other causes).
Medication adherence | For the duration of the study: 3 months
  Reported as the number of patients self-reporting "all assigned medications were taken" "missing at least one dose of study medication", or "not able to take all of the study medications" out of the total number of medication compliance assessments done respectively.
Quality-adjusted life years (QALYs) gained | For the duration of the study: 3 months
  We will measure health utility values using the EuroQoL-5D-5L 51 at baseline, 2 week (± 7 days), and 90 days (+14 days). We will model the prognosis of a cohort of patients receiving rivaroxaban as a baseline against the potential impact of apixaban. The results will be presented as incremental cost per QALY gained, incremental costs per one CRB cases prevented, and incremental cost per one life year saved.
Incremental cost-effectiveness ratio | For the duration of the study: 3 months
  Incremental cost-effectiveness ratios including cost per one CRB case prevented, cost per one life year saved, cost per one quality-adjusted life year (QALY) gained, which will be analyzed as part of the health economic analysis plan.
Impact of verbal consent on patient participation in comparison with participants from sites using written informed consent | For the duration of the study: 3 months
  Impact of verbal consent on patient participation in comparison with participants from sites using written informed consent. Due to the qualitative nature of this outcome, it will be presented descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Lana Castellucci, MD, FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (19):
- The University of Sydney, Darlington, New South Wales, Australia
- Canada (17):
  - University of Calgary, Calgary, Alberta
  - Alberta Health Sciences, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Center, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - UHN - Toronto General Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - St. Mary's Hospital, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec
- The Royal College of Surgeons in Ireland/Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No